CLINICAL TRIAL: NCT06971484
Title: Comparative Bioavailability of Crystalline and Regular Glucosamine Sulfate: A Randomized Crossover Study in Healthy Adults
Brief Title: Glucosamine Sulfate Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-11-002GS
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Bioavailability and Pharmacokinetics
Keywords: glucosamine; crystalline; pharmacokinetics; bioavailability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalline glucosamine sulfate (Experimental): Participants receive their treatment of crystalline glucosamine sulfate at a total dose of 1500 mg of glucosamine sulfate. Treatments are consumed with a glass of water followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at different time points up to 24 hours post-dose. A washout period of 1 week between each treatment is used.
  Interventions: Dietary Supplement: Crystalline glucosamine sulfate
- Regular glucosamine sulfate (Experimental): Participants receive their treatment of regular glucosamine sulfate at a total dose of 1500 mg of glucosamine sulfate. Treatments are consumed with a glass of water followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at different time points up to 24 hours post-dose. A washout period of 1 week between each treatment is used.
  Interventions: Dietary Supplement: Regular glucosamine sulfate

INTERVENTIONS:
Dietary Supplement: Crystalline glucosamine sulfate — A maximum single dose of 1500mg of glucosamine sulfate in a caplet.
  Arms: Crystalline glucosamine sulfate
Dietary Supplement: Regular glucosamine sulfate — A maximum single dose of 1500mg of glucosamine sulfate in hard gel capsules.
  Arms: Regular glucosamine sulfate

SUMMARY:
This study aims to compare the pharmacokinetics and bioavailability of crystalline glucosamine sulfate and regular glucosamine sulfate using a double-blind, randomized, crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 21- 65 years
* Healthy, good physical condition
* Voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* Serious acute or chronic diseases e.g. liver, kidney, or gastrointestinal diseases
* Use of medications affecting glucosamine metabolism
* Known allergies to shellfish or glucosamine
* Pregnancy or breastfeeding
* Participation in another investigational study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
AUC: the area under the concentration-time curve | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested glucosamine sulfate in healthy adult volunteers and compare the Area under the plasma concentration versus time curve (AUC) with that of other capsules containing glucosamine sulfate.
Cmax: maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested glucosamine sulfate in healthy adult volunteers and compare the peak plasma concentration (Cmax) with that of other capsules containing glucosamine sulfate.
Tmax: the time point of maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested glucosamine sulfate in healthy adult volunteers and compare the time point of maximum plasma concentration (Tmax) with that of other capsules containing glucosamine sulfate.

CONTACTS AND LOCATIONS:
Locations (1):
- ISURA, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No